CLINICAL TRIAL: NCT02055170
Title: Neoadjuvant Finasteride for Patients With Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to improve on poor accrual to study.
Sponsor: CancerCare Manitoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLC001
Record Dates: First submitted 2014-02-02; First posted 2014-02-05 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Finasteride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- finasteride (Experimental): finasteride 5mg po od from study entry to date of surgery
  Interventions: Drug: finasteride 5mg oral daily

INTERVENTIONS:
Drug: finasteride 5mg oral daily

SUMMARY:
The purpose of this study is to study the effect of hormone therapies (androgen pathway modification) on the outcomes of patients with lung cancer. This information may be of benefit for future treatment strategies, prevention and control.

In this study, the protein where testosterone binds, called the androgen receptor (AR), will be measured in samples from the patient's biopsy and surgical tumor samples. The investigators will look at a marker of how fast the cancer is growing (Ki67) before using finasteride from your biopsy specimen. Finasteride will be taken from the day of consent until the day of the patient's surgery. This marker will be measured again after using finasteride from the surgical specimen. The investigators will be looking for a decrease in the Ki67 from the patient's biopsy specimen to the surgical specimen as an indicator that this medication is blocking tumour growth.

ELIGIBILITY:
Inclusion Criteria:

* male
* age >18
* biopsy-proven non-small cell lung cancer
* surgical intervention planned

Exclusion Criteria:

* current use of 5-alpha reductase inhibitor
* previous diagnosis of prostate cancer
* previous hypersensitivity to 5-alpha reductase inhibitor

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-06; Primary Completion 2018-03-27 (Actual); Study Completion 2018-03-27 (Actual)

PRIMARY OUTCOMES:
Change in proliferation | Original biopsy to surgical specimen (approx 6 weeks)
  Patients will be followed from time of consent (around the time of consultation with a Thoracic Surgeon) to date of surgery (on average, approximately 4-6 weeks following Thoracic Surgeon consultation).

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences Centre, Winnipeg, Manitoba, Canada